CLINICAL TRIAL: NCT06382155
Title: A Phase 2, Randomized, Controlled, Multicenter Study of Vosoritide in Children with Idiopathic Short Stature
Brief Title: A Phase 2 Study of Vosoritide in Children with Idiopathic Short Stature
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-210
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Short Stature
MeSH Terms: interventions — vosoritide; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Vosoritide Dose 1 - Low Dose (Experimental): Vosoritide Dose 1 daily injection
  Interventions: Drug: Vosoritide Injection
- Vosoritide Dose 2 - Medium Dose (Experimental): Vosoritide Dose 2 daily injection
  Interventions: Drug: Vosoritide Injection
- Vosoritide Dose 3 - High Dose (Experimental): Vosoritide Dose 3 daily injection
  Interventions: Drug: Vosoritide Injection
- Placebo (Placebo Comparator): Placebo daily injection
  Interventions: Drug: Placebo
- Human Growth Hormone (Active Comparator): hGH daily injection
  Interventions: Drug: Human Growth Hormone

INTERVENTIONS:
Drug: Vosoritide Injection — Experimental Drug Lyophilized powder for reconstitution
  Arms: Vosoritide Dose 1 - Low Dose; Vosoritide Dose 2 - Medium Dose; Vosoritide Dose 3 - High Dose
Drug: Human Growth Hormone — Commercial product containing somatotropin
  Arms: Human Growth Hormone
Drug: Placebo — Lyophilized powder for reconstitution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate i) the effect of multiple doses of vosoritide and ii) the effect of the therapeutic dose of vosoritide compared to human growth hormone (hGH), in children with idiopathic short stature (ISS).

DETAILED DESCRIPTION:
Following a minimum 6 month observational period in which baseline growth is assessed, participants in the vosoritide and placebo groups will complete a minimum of 6 months of randomized treatment (maximum of 6 months of placebo treatment), followed by open-label treatment with vosoritide until they reach near-final adult height, or at least 16 years of age for females or 18 years of age for males, whichever comes later. Participants randomized to the hGH group will receive open-label hGH for a minimum of 4 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Height assessment corresponding to a height Z-score of ≤ -2.25 SDs in reference to the general population of the same age and sex, as calculated using the Centers for Disease Control and Prevention (CDC) growth charts
2. Tanner Stage 1, at time of signing the ICF (unless too young to stage).

Key Exclusions:

1. Known chromosomal imbalance or genetic variant causing short stature syndrome, including but not limited to Laron syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, Turner syndrome, disproportionate skeletal dysplasias, abnormal SHOX gene analysis, or Rasopathy (including Noonan syndrome)
2. Previous treatment with a growth promoting agent

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participants must be ≥ 3 years old, and < 10 years old (female) or < 11 years old (males) at the time of signing the informed consent form (ICF).
Enrollment: 100 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Annualized Growth Velocity (AGV) | At 6 months
Change from baseline in height | At 4 years
Change from baseline in height Z-score | At 4 years

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Until the end of the study, up to 15 years
Change from baseline in AGV Z-score (average stature reference) | At 6 months
Change from baseline in height | Every 6 months through the end of study, up to 15 years
Change from baseline in height Z score | Every 6 months through the end of study, up to 15 years
Change from baseline at prespecified timepoints in urine cyclic guanine monophosphate (cGMP) | Every 6 months through the end of study, up to 15 years
Change from baseline at pre-specified timepoints in serum collagen X marker (CXM) | Every 6 months through the end of study, up to 15 years
Change from baseline in bone age minus chronological age at pre-specified timepoints | Every 6 months through the end of study, up to 15 years
Change from baseline in total body (less head) bone mineral density (BMD) Z-score | Every 6 months through the end of study, up to 15 years
Change from baseline in lumbar spine BMD Z-score | Every 6 months through the end of study, up to 15 years
Change from baseline in total body (less head) bone mineral content (BMC) | Every 6 months through the end of study, up to 15 years
Change from baseline in lumbar spine BMC | Every 6 months through the end of study, up to 15 years
Maximum concentration (Cmax) of vosoritide in plasma | Every 6 months through the end of study, up to 15 years
Area under the plasma vosoritide concentration time-curve from time 0 to infinity (AUC0-∞) | Every 6 months through the end of study, up to 15 years
Area under the plasma vosoritide concentration time-curve from time 0 to the last measurable concentration (AUC0-t) | Every 6 months through the end of study, up to 15 years
Elimination half-life of vosoritide (t½) | Every 6 months through the end of study, up to 15 years
Apparent clearance of vosoritide | Every 6 months through the end of study, up to 15 years
Apparent volume of distribution of vosoritide based upon the terminal phase (Vz/F) | Every 6 months through the end of study, up to 15 years
Time vosoritide is present at maximum concentration (Tmax) | Every 6 months through the end of study, up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director MD, Study Director — BioMarin Pharmaceutical
Locations (8):
- United States (8):
  - Center Of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Lundquist Institute for Biomedical Innovation (LA BioMed), Torrance, California
  - Nemours Children's Health System - Corporate Headquarters, Pensacola, Florida
  - Centricity Research, Columbus, Georgia
  - St. Luke's Children's Endocrinology, Boise, Idaho
  - Rocky Mountain Clinical Research - Idaho Falls, Idaho Falls, Idaho
  - UBMD Pediatrics, Buffalo, New York
  - Children's Hospital at Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided